CLINICAL TRIAL: NCT04364412
Title: Acute Lower gastroIntestinal BleedIng (ALIBI Study): a Multicentre Prospective, Cohort Study
Brief Title: Acute Lower gastroIntestinal BleedIng (ALIBI Study) in Italy
Acronym: ALIBI
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Head of Gastroenterology Department, Valduce Hospital
Other Study IDs: 70/2018
Record Dates: First submitted 2020-04-06; First posted 2020-04-28 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Lower GI Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Unlike upper GI bleeding, for LGIB there is still a paucity of data on clinical presentation, patient characteristics, pathways of care and outcomes for LGIB patients. In-hospital mortality ranges from 1.2% to 8.8% (2-4), according to retrospective studies, but data from prospective series are still limited (5).

Present multicentre, prospective, observational study was designed to explore these areas, to assess variations in practice management and to identify factors associated with patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with acute lower GI bleeding

Exclusion Criteria:

* age below 18 years
* bleeding patients with an upper GI source

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive, unselected outpatients acutely admitted for LGIB or developing LGIB during hospital stay (inpatients) were eligible for inclusion if they fulfilled the following criteria: i) age > 18 years; ii) recent (< 3 days) onset of overt bleeding with bright or dark blood or clots per rectum or melaena without hematemesis
Sampling Method: Probability Sample
Enrollment: 1198 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Mortality rate in patients admitted for acute lower GI bleeding | 4 weeks
  Number of deaths among the study cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, Italy

REFERENCES:
- [Derived] Radaelli F, Frazzoni L, Repici A, Rondonotti E, Mussetto A, Feletti V, Spada C, Manes G, Segato S, Grassi E, Musso A, Di Giulio E, Coluccio C, Manno M, De Nucci G, Festa V, Di Leo A, Marini M, Ferraris L, Feliziani M, Amato A, Soriani P, Del Bono C, Paggi S, Hassan C, Fuccio L. Clinical management and patient outcomes of acute lower gastrointestinal bleeding. A multicenter, prospective, cohort study. Dig Liver Dis. 2021 Sep;53(9):1141-1147. doi: 10.1016/j.dld.2021.01.002. Epub 2021 Jan 25. PMID 33509737